CLINICAL TRIAL: NCT02178579
Title: Prospective Observation of Cardiac Safety With Proteasome Inhibition
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 140404
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure; Multiple Myeloma
Keywords: Heart Failure; Cardiac Toxicity; Multiple Myeloma; Bortezomib; Carfilzomib
MeSH Terms: conditions — Heart Failure; Multiple Myeloma; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample banked for future research.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multiple Myeloma (MM) treatment with bortezomib: No intervention planned.
- Multiple Myeloma (MM) treatment with carfilzomib: No intervention planned.

SUMMARY:
The purpose of this study is to better define and understand potential cardiac toxicities of proteasome inhibitors and to understand optimal management strategies to treat and prevent cardiovascular events.

DETAILED DESCRIPTION:
Cancer treatments, using proteasome inhibitors, have the potential in induce cardiac toxicities including heart failure (HF), hypertension, arrhythmias and ischemic heart disease. While the presence of cardiac events may be a class effect of proteasome inhibitors (PI), the effect may be more profound with the irreversible inhibition of carfilzomib compared with reversible inhibition with bortezomib. Data available from currently published clinical trials may be inadequate to fully understand the incidence and severity of cardiac injury in patients treated with proteasome inhibitors because the trials were not designed to fully assess cardiac events. The purpose of this study is to better define and understand potential cardiac toxicity and begin to understand optimal management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed multiple myeloma at any time-point in treatment course and planning to start a proteasome inhibitor-based therapy as part of standard care
* Received at least one prior line of therapy for multiple myeloma (induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as one line of therapy)
* Males and females ≥ 18 years of age
* Able to provide written informed consent in accordance with federal, local, and institutional guidelines

Exclusion Criteria:

* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Known or suspected AL amyloidosis, secondary amyloidosis or cardiac amyloidosis
* Plasma cell leukemia (> 2.0 × 109/L circulating plasma cells by standard differential)
* Waldenström Macroglobulinemia
* Myelodysplastic syndrome
* History of MI within the last 3 months
* Symptomatic unstable cardiac arrhythmia requiring treatment in the past 3 months
* Class 3 or 4 New York Heart Association Heart Failure in the past 3 months
* Any other clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma patients being treated with bortezomib or carfilzomib, per oncology physician decision.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Frequency of cardiac events of patients receiving PIs for MM. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Cornell, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - University of Pennsylvania/Smilow Center for Translational Research, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.

REFERENCES:
- [Derived] Cornell RF, Ky B, Weiss BM, Dahm CN, Gupta DK, Du L, Carver JR, Cohen AD, Engelhardt BG, Garfall AL, Goodman SA, Harrell SL, Kassim AA, Jadhav T, Jagasia M, Moslehi J, O'Quinn R, Savona MR, Slosky D, Smith A, Stadtmauer EA, Vogl DT, Waxman A, Lenihan D. Prospective Study of Cardiac Events During Proteasome Inhibitor Therapy for Relapsed Multiple Myeloma. J Clin Oncol. 2019 Aug 1;37(22):1946-1955. doi: 10.1200/JCO.19.00231. Epub 2019 Jun 12. PMID 31188726